CLINICAL TRIAL: NCT04434378
Title: The Use of Tamsulosin to Prevent Postoperative Urinary Retention in Laparoscopic Inguinal Hernia Repair: A Randomized Double-Blind Placebo-Controlled Study
Brief Title: Tamsulosin to Prevent Postoperative Urinary Retention in Laparoscopic Inguinal Hernia Repair
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Significant difference not reached on interim analysis
Sponsor: Jewish Hospital, Cincinnati, Ohio (Other)
Responsible Party: Principal Investigator, Michael Caparelli, Resident, Jewish Hospital, Cincinnati, Ohio
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17-19
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Post Operative Urinary Retention
Keywords: laparoscopic inguinal hernia repair; tamsulosin
MeSH Terms: interventions — Tamsulosin

STUDY DESIGN:
Intervention Model Description: One group will be randomized to tamsulosin and the second group randomized to placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients undergoing laparoscopic inguinal hernia repair will randomized to one dose of placebo in the preoperative holding area 2 hours before surgery.
  Interventions: Drug: Placebo
- Interventional (Experimental): Patients undergoing laparoscopic inguinal hernia repair will be randomized to one dose of 0.4 mg tamsulosin in the preoperative holding area 2 hours before surgery.
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Drug: Tamsulosin — 0.4 mg tamsulosin will be given to a randomized group of patients
  Arms: Interventional
Drug: Placebo — placebo will be given to a randomized group of patients
  Arms: Placebo

SUMMARY:
To investigate the effect of tamsulosin on the development of post-operative urinary retention (PUR) after elective laparoscopic inguinal hernia repair (LIHR). This will be accomplished by administering a pre-operative dose of tamsulosin. The primary outcome is the rate of urinary retention necessitating straight catheterization or insertion of foley catheter prior to discharge.

DETAILED DESCRIPTION:
Patients who are scheduled for elective laparoscopic inguinal hernia repair will be consented in the office by the attending physician. An order will be placed during surgery scheduling for tamsulosin with instruction to administer one dose in the preoperative holding area on the day of surgery. The Jewish hospital pharmacy will be responsible for providing randomization and placebo medications for double blinding effect. PUR will be tracked on the basis of urinary catheterization performed prior to hospital discharge. Criteria for catheterization include: i) Inability to urinate within 6 hours post-operatively, and bladder scan showing >400 mL. ii) Inability to urinate at any time postoperatively with symptoms of urinary retention (i.e. urgency, bladder discomfort). Women of childbearing age will need to have a confirmed negative urine or serum pregnancy test prior to surgery. This will be completed on arrival to the preoperative holding area.

To detect the difference between the treated group and control group with a significant alpha (0.5) and power (80%), at least 178 patients will be needed in each group. This was generated using the Pearson Chi-square test for Two proportions.

This study will be conducted in the hospital setting at a single institution. Patients will be consented for the study in the pre-admission holding area and followed until discharged from the post anesthesia care unit.

ELIGIBILITY:
Inclusion Criteria:

1. All patients undergoing elective laparoscopic inguinal hernia repair, unilateral or bilateral.
2. ≥18 years of age.
3. Patients must leave the operating room without at indwelling urinary catheter.

Exclusion Criteria:

1. History of neurogenic bladder requiring routine intermittent catheterization
2. Emergent laparoscopic hernia repair.
3. Elective laparoscopic hernia repair in conjuncture with an additional operation (e.g. nephrectomy, pelvic surgery) that requires the patient to have a planned, indwelling urinary catheter in the postoperative period.
4. Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative urinary retention. | Within 24 hours of surgery
  Patients undergoing laparoscopic inguinal hernia repair will be assessed for postoperative urinary retention in the post anesthesia care unit. Postoperative urinary retention will be tracked on the basis of urinary catheterization performed prior to hospital discharge. Criteria for catheterization include: i) Inability to urinate within 6 hours post-operatively, and bladder scan showing >400 mL. ii) Inability to urinate at any time postoperatively with symptoms of urinary retention (i.e. urgency, bladder discomfort).

SECONDARY OUTCOMES:
Incidence of risk factors for postoperative urinary retention in patients undergoing laparoscopic inguinal hernia repair. | within 24 hours of surgery
  Retrospective chart review will be utilized to asses the incidence of risk factors of postoperative urinary retention in patients undergoing laparoscopic inguinal hernia repair. Risk factors including age >60, total IV fluids, length of procedure, opioid use, bilateral vs unilateral repair, BMI >30, diabetes mellitus, coronary artery disease, and benign prostatic hyperplasia will be assessed. These risk factors will then undergo statistical analysis to determine if they are associated with postoperative urinary retention.

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garg P, Rajagopal M, Varghese V, Ismail M. Laparoscopic total extraperitoneal inguinal hernia repair with nonfixation of the mesh for 1,692 hernias. Surg Endosc. 2009 Jun;23(6):1241-5. doi: 10.1007/s00464-008-0137-0. Epub 2008 Sep 24. PMID 18813990
- [Background] Mohammadi-Fallah M, Hamedanchi S, Tayyebi-Azar A. Preventive effect of tamsulosin on postoperative urinary retention. Korean J Urol. 2012 Jun;53(6):419-23. doi: 10.4111/kju.2012.53.6.419. Epub 2012 Jun 19. PMID 22741052
- [Background] Shaw MK, Pahari H. The role of peri-operative use of alpha-blocker in preventing lower urinary tract symptoms in high risk patients of urinary retention undergoing inguinal hernia repair in males above 50 years. J Indian Med Assoc. 2014 Jan;112(1):13-4, 16. PMID 25935942
- [Background] Sivasankaran MV, Pham T, Divino CM. Incidence and risk factors for urinary retention following laparoscopic inguinal hernia repair. Am J Surg. 2014 Feb;207(2):288-92. doi: 10.1016/j.amjsurg.2013.06.005. Epub 2013 Nov 5. PMID 24200291